CLINICAL TRIAL: NCT02571075
Title: A Randomized, Single-blind, Prospective Trial of Auricular Acupuncture for the Reduction of Post-operative Tonsillectomy Pain in Adults
Brief Title: Battlefield Auricular Acupuncture During Adult Tonsillectomies and Effect of Post op Pain and Nausea
Acronym: BFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 381600
Record Dates: First submitted 2015-10-02; First posted 2015-10-08 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Tonsillitis
Keywords: auricular; acupuncture; pain
MeSH Terms: conditions — Tonsillitis; Pain | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 - Receives auricular acupuncture (Experimental): Receives "Battlefield Acupuncture" (BFA) as soon a anesthesia is initiated and needles removed right before they are extubated and awakened.
  Interventions: Other: Auricular acupuncture
- Group 2 don't receive anything (No Intervention): They do not receive any any acupuncture only standard of care.

INTERVENTIONS:
Other: Auricular acupuncture — The ear will be cleaned with alcohol prior to insertion of the needles. Five sterile, single-use, gold needles will be placed in each ear according to the figure below. The needles penetrate about a millimeter (or 4/100ths of an inch) into the skin.
  Other Names: "Battlefield Acupuncture" BFA
  Arms: Group 1 - Receives auricular acupuncture

SUMMARY:
The purpose of this study is to determine if auricular acupuncture significantly reduces post-operative pain in comparison to the standard of care. Post-operative pain score will be collected by subject self-report of pain according to the Numerical Rating Scale (NRS) (0= no pain, 10 = worst imaginable pain) up to 10 days post-operation.

DETAILED DESCRIPTION:
DESIGN:

Design type: Prospective, randomized control trial Sample

* Description of the population: All adults, greater than or equal to 18 years, undergoing a tonsillectomy with or without adenoidectomy at Womack Army Medical Center are eligible for participation in the study.
* Sample Size: 100 subjects. A target of 45 subjects per group for a total of 90 subjects, and accounting for a 10 percent drop out rate. In Fiscal Year 12, 92 tonsilectomies in patients over the age of 12 were performed at Womack Army Medical Center. Therefore, the investigators anticipate the study will take up to 4 years to enroll 100 adult subjects.
* Power Analysis: Under the assumption of a linear time by treatment interaction, assuming subject-level randomization, five time-points, power of 80 percent, a Type I error rate of 5 per cent and no attrition, to detect a 1.6 difference in pain score requires a total sample size of 90 subjects or 45 per treatment arm.

ELIGIBILITY:
Inclusion Criteria

* All adults eighteen years of age or older having a tonsillectomy with or without adenoidectomy
* Anesthesiologist classification one to three

Exclusion Criteria

* Chronic pain syndromes or pain symptoms lasting greater than three months or taking opioids on a daily basis for greater than four months
* Anesthesiologist classification four
* Prior neck or throat surgery
* Allergy to gold

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-11; Primary Completion 2017-06-08 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Plunkett, MD, Principal Investigator — Womack Army Medical Center Fort Bragg
Locations (1):
- Womack Army Medical Center, Fort Bragg, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 - Receives Auricular Acupuncture | Group 2 Don't Receive Anything
Started | 45 | 50
Completed | 25 | 26
Not Completed | 20 | 24
Not completed — Lost to Follow-up | 20 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Receives Auricular Acupuncture | Group 2 Don't Receive Anything | Total
Number analyzed (Participants) | 45 | 50 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 50 | 95
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 25 [22 to 30] | 26 [22 to 29] | 25 [22 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 51
  Male | 21 | 23 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 2 | 1 | 3
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 9 | 5 | 14
  Race: White | 27 | 32 | 59
  Race: More than one race | 0 | 0 | 0
  Race: Unknown or Not Reported | 7 | 12 | 19
Region of Enrollment [Number; unit: participants]
  United States | 45 | 50 | 95

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores
Description: Pain scores will be collected daily during the post op period in the recovery room using a numbers scale with faces; specifically the Wong-Baker FACES® Pain Rating Scale where 10 is described as worst possible and 0 is No pain. This was recorded by the participant at home using the same type scale and this was is provided to them. The Hypothesis is that subjects receiving intraoperative auricular acupuncture during a tonsillectomy will have statistically significantly less post-operative pain scores compared to those that do not.
Time Frame: 10 days after the procedure.
Population: Only a 50 % diary return completing the full 10 day diary data but had the full inpatient data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 - Receives Auricular Acupuncture | Group 2 Don't Receive Anything
Number analyzed (Participants) | 45 | 50
units on a scale
  Pain at discharge: number analyzed (Participants) | 44 | 49
  Pain at discharge | 1.3 (1.6) | 1.4 (1.6)
  Pain at 6 hours post discharge: number analyzed (Participants) | 23 | 23
  Pain at 6 hours post discharge | 5.1 (1.6) | 5.9 (2.1)
  12 hours post discharge: number analyzed (Participants) | 22 | 50
  12 hours post discharge | 5.5 (1.9) | 6.4 (1.9)
  18hrs post discharge: number analyzed (Participants) | 22 | 24
  18hrs post discharge | 5.4 (1.7) | 6.4 (1.6)
  24 hrs post discharge: number analyzed (Participants) | 24 | 24
  24 hrs post discharge | 5.3 (2.1) | 6.0 (2.1)
  day 2 of discharge: number analyzed (Participants) | 24 | 26
  day 2 of discharge | 6.1 (1.9) | 6.5 (2.0)
  day 3 of discharge: number analyzed (Participants) | 23 | 26
  day 3 of discharge | 5.8 (2.1) | 6.4 (2.2)
  day 4 of discharge: number analyzed (Participants) | 23 | 25
  day 4 of discharge | 5.6 (1.9) | 5.6 (1.9)
  day 5 of discharge: number analyzed (Participants) | 22 | 25
  day 5 of discharge | 5.5 (2.2) | 6.3 (1.9)
  day 6 of discharge: number analyzed (Participants) | 22 | 25
  day 6 of discharge | 5.5 (2.3) | 6.2 (2.2)
  day 7 of discharge: number analyzed (Participants) | 22 | 25
  day 7 of discharge | 5.3 (2.3) | 5.3 (2.3)
  day 8 of discharge: number analyzed (Participants) | 22 | 25
  day 8 of discharge | 4.6 (2.3) | 5.5 (2.3)
  day 9 of discharge: number analyzed (Participants) | 18 | 25
  day 9 of discharge | 4.4 (2.5) | 4.7 (2.1)
  Day 10 of discharge: number analyzed (Participants) | 17 | 22
  Day 10 of discharge | 3.6 (2.1) | 3.9 (2.2)

2. Primary Outcome: The Morphine Equivalent of Opioid Use
Description: The intraoperative and recovery room morphine equivalents will be calculated and upon diary return what use is recorded by the patient will be done as well. The participant is instructed to write down the type and amount they take throughout that time period.
Time Frame: Intraoperative to 10 days post operative utilizing the Johns Hopkins Opioid conversion system.
Population: Some results based on 10 day diary return but inpatient data available on all subjects
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group 1 - Receives Auricular Acupuncture | Group 2 Don't Receive Anything
Number analyzed (Participants) | 45 | 50
mg
  Oral morphine equivalent in OR in mg | 63.8 (2407) | 70.5 (24.0)
  oral morphine equivalent in PACU in mg | 9.1 (20.0) | 7.4 (10.9)
  oral morphine equivalent in mg 10 days post discha: number analyzed (Participants) | 23 | 26
  oral morphine equivalent in mg 10 days post discha | 257.3 (341.7) | 295.7 (257.8)
  oral morphine equivalent total OR+ PACU+Home: number analyzed (Participants) | 23 | 26
  oral morphine equivalent total OR+ PACU+Home | 334.3 (339.4) | 376.2 (254.3)

3. Secondary Outcome: Return to Diet
Description: Subjects will record on their diary the date they returned to a regular diet (defined to them what is regular for them)
Time Frame: Within 10 days post operatively
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1 - Receives Auricular Acupuncture | Group 2 Don't Receive Anything
Number analyzed (Participants) | 17 | 22
days | 10 (1.9) | 10 (1.9)

4. Secondary Outcome: Number of Participants With Nausea Post Operatively
Description: It will be documented yes or no if the participant voiced any complaint of nausea while in recovery.
Time Frame: 1-3 hours postoperativey
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Receives Auricular Acupuncture | Group 2 Don't Receive Anything
Number analyzed (Participants) | 45 | 50
Participants | 6 | 3

5. Secondary Outcome: Number of Participants With Nausea Post Operatively
Description: It will be documented yes or no if the participant had any emesis while in recovery prior to discharge home.
Time Frame: 1-3 hours post operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Receives Auricular Acupuncture | Group 2 Don't Receive Anything
Number analyzed (Participants) | 45 | 50
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 3 years from first enrolled to final participant
Arm/Group | Group 1 - Receives Auricular Acupuncture | Group 2 Don't Receive Anything
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/50
Other Adverse Events (participants affected / at risk) | 2/45 | 3/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Receives Auricular Acupuncture (N=45) | Group 2 Don't Receive Anything (N=50)
Emergency room visit (General disorders) | 2 (2) | 3 (3) — bleeding

LIMITATIONS AND CAVEATS:
Of the 95 enrolled there was only a 50% diary return of the 10 day diaries and not all of those were complete.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT02571075/Prot_SAP_000.pdf